CLINICAL TRIAL: NCT02152189
Title: Screening for Fabry Disease in a Pediatric Population at Risk
Status: Completed | Type: Observational
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Markus Ries, MD PhD MHSc FCP, Professor, University Hospital Heidelberg
Other Study IDs: Fabry screening 02202014; S-084/2014 (Other: IRB Heidelberg)
Record Dates: First submitted 2014-05-22; First posted 2014-06-02 (Estimated); Last update posted 2017-12-13 (Actual); Status verified 2017-12

CONDITIONS: Chronic Pain in the Extremities; Chronic Abdominal Pain; Fabry Disease
MeSH Terms: conditions — Fabry Disease | interventions — Mass Screening

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Screening population
  Interventions: Other: Screening for Fabry disease

INTERVENTIONS:
Other: Screening for Fabry disease

SUMMARY:
The purpose of this study is to assess the frequency of Fabry disease in children with chronic abdominal pain or chronic pain in the extremities

ELIGIBILITY:
Inclusion Criteria:

* Age below 18 years
* One of the following criteria:

  * Diagnosis or suspicion of a rheumatological disorder with recurrent complaints for more than 6 months
  * Chronic, recurrent abdominal pain for more than 6 months
* Planned blood sample for routine diagnostics
* Written informed consent

Exclusion Criteria:

- Patient and/or the patient's parent(s) or legal guardian(s) are unable to understand the nature, scope, and possible consequences of the screening.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with rheumatological disorders or chronic abdominal pain
Sampling Method: Probability Sample
Enrollment: 1422 (Actual)
Dates: Start 2014-05; Primary Completion 2017-05 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Prevalence of Fabry disease | day 1

SECONDARY OUTCOMES:
Prevalence of Fabry disease in predefined sub-populations | day 1

CONTACTS AND LOCATIONS:
Locations (1):
- Zentrum für Kinder- und Jugendmedizin, Heidelberg, Germany

REFERENCES:
- [Background] Ries M, Gupta S, Moore DF, Sachdev V, Quirk JM, Murray GJ, Rosing DR, Robinson C, Schaefer E, Gal A, Dambrosia JM, Garman SC, Brady RO, Schiffmann R. Pediatric Fabry disease. Pediatrics. 2005 Mar;115(3):e344-55. doi: 10.1542/peds.2004-1678. Epub 2005 Feb 15. PMID 15713906
- [Derived] Kastner B, Behre S, Lutz N, Burger F, Luntz S, Hinderhofer K, Bendszus M, Hoffmann GF, Ries M. Clinical Research in Vulnerable Populations: Variability and Focus of Institutional Review Boards' Responses. PLoS One. 2015 Aug 14;10(8):e0135997. doi: 10.1371/journal.pone.0135997. eCollection 2015. PMID 26275228